CLINICAL TRIAL: NCT06968468
Title: Resilient Together-ALS (RT-ALS): A Dyadic Mind-body Meaning Intervention for People With ALS and Their Informal Care-partners
Brief Title: Resiliency Intervention for Patients With ALS and Their Care-Partners
Acronym: RT-ALS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christina Rush, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001058
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Emotional Distress
Keywords: Amyotrophic Lateral Sclerosis; ALS; Caregiving; Coping
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT-ALS Intervention (Experimental): Dyads will participate in 6 30-45-minute skills based sessions. A clinical psychologist will deliver all sessions. The main intervention goal is to provide dyads with coping and resiliency skills and resources to reduce emotional distress, prevent chronic distress, and preserve quality of life for both dyad members as ALS progresses.
  Interventions: Behavioral: Resilient Together ALS

INTERVENTIONS:
Behavioral: Resilient Together ALS — This intervention will teach resiliency and coping skills (mindfulness, meaning making, etc) to dyads soon after ALS diagnosis in order to manage distress associated with an ALS diagnosis. These sessions will take place over Zoom with both the person diagnosed with ALS and their primary informal caregiver.

SUMMARY:
The purpose of this study is to pilot a resiliency and coping intervention for persons recently diagnosed with Amyotrophic Lateral Sclerosis (ALS) and their primary informal caregivers. The data investigators gather in this study will be used to further refine our intervention.

DETAILED DESCRIPTION:
The goal of this study to refine our proposed intervention Resilient Together ALS (RT-ALS) through an open pilot. The investigators will deliver an open pilot of the intervention (N= up to10 dyads; up to 20 participants total) to evaluate initial feasibility and acceptability using exit interviews and pre-post assessments.

The open pilot will take place over Zoom, with participants recruited from the Massachusetts General Hospital's Sean M. Healey and AMG Center for ALS. Study clinicians will deliver 6, 30-45 minute sessions over Zoom. All participants will complete measures at baseline and after completion of the program (6 weeks). At the completion of the program, participants will engage in an exit interview where they will provide feedback on the intervention.

ELIGIBILITY:
Inclusion Criteria for patient with ALS:

* recent (within ~2 months) of first appointment at Healey Center for diagnosis of ALS documented in Epic (based on recommendations from neurologists)
* ability to understand the study and research protocol as determined by a standardized teach-back method of assessment
* ability to communicate by writing, speaking, or assistive communication device

Inclusion Criteria for dyad:

* English speaking adults
* dyad lives together
* at least one partner endorses clinically significant emotional distress during screening (>7 on either subscale of the HADS)

Exclusion Criteria:

* patient with ALS with comorbid terminal diagnosis or severe mental health disorder that limits ability to participate (by self-report, as determined by our clinical team);
* cognitive disorder that limits ability to participate (per neurologist)
* inability or unwillingness to use live video technology (will teach any dyads who have low technology literacy how to use live video technology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-05-13 (Estimated); Primary Completion 2027-02-13 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | 0 weeks
  Percentage of eligible ALS patient-caregiver dyads that participate in the intervention (>70% acceptable; >80% excellent).
Data Collection Feasibility | Pre-test (0 weeks) to Post-test (6 weeks)
  Percentage of dyads with no missing measures (>70% acceptable; >80% excellent)
Adherence Feasibility | 6 weeks
  Percentage of RT-ALS dyads that complete 4/6 sessions (>70% acceptable; >80% excellent)
Therapist Fidelity Feasibility | 6 weeks
  Percentage of adherence checklists completed; percentage of selected sessions (20%) with 100% adherence Fidelity Checks (>70% acceptable; >80% excellent).
Treatment Satisfaction | 6 weeks
  Percentage of dyads who score above the midpoint on Client Satisfaction Questionnaire (> 70% acceptable; > 80% excellent)
Credibility and Expectancy | Pre-test (0 weeks)
  Percentage of dyads who score above midpoint on the Credibility/Expectancy Questionnaire (> 70% acceptable; > 80% excellent)
Adverse Events | 6 weeks
  None or minimal adverse events

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Pre-test (0 weeks) to Post-test (6 weeks)
  Report of emotional distress at baseline and post-test as measured by the Hospital Anxiety and Depression Scale (HADS). Minimum score: 0 Maximum score: 21 for both the Anxiety and Depression sub-scales. Higher scores indicate higher levels of reported anxiety and depression.
The World Health Organization Quality of Life abbreviated (WHOQOL-BREF) | Pre-test (0 weeks) to Post-test (6 weeks)
  Quality of life of RT-ALS dyads reported at both baseline and post-test as measured by the World Health Organization Quality of Life - abbreviated measure (WHOQOL-BREF). Maximum score: 20 Minimum score: 4 on each domain. Higher scores indicate higher quality of life.
Cognitive and Affective Mindfulness Scale (CAMS) | Pre-test (0 weeks) to Post-test (6 weeks)
  The Cognitive and Affective Mindfulness Scale (CAMS) measures dispositional mindfulness, higher values reflect higher levels of mindfulness. Maximum score: 48 Minimum score: 12.
Measure of Current Status Part A (MOCS-A) | Pre-test (0 weeks) to Post-test (6 weeks)
  Assesses ability to engage in a series of healthy coping skills (e.g., relaxation, social support, adaptive thinking). Maximum score: 52 Minimum score: 0; higher scores indicate a greater perceived ability to employ adaptive coping strategies.
Multidimensional Scale of Perceived Social Support (MSPSS) | Pre-test (0 weeks) to Post-test (6 weeks)
  A measure of perceived social support. Higher scores indicate greater perceived social support. Minimum score: 1 Maximum score: 7.
Dyadic Coping Inventory (DCI) | Pre-test (0 weeks) to Post-test (6 weeks)
  Assesses self-reported coping behaviors when dyad faces stressors. Higher scores reflect more adaptive coping. Maximum score: 35 Minimum score: 1.
The Meaning in Life Questionnaire (MLQ) | Pre-test (0 weeks) to Post-test (6 weeks)
  A measure of sense of meaning and purpose in life. A higher score on the presence of meaning items indicates higher presence of meaning. A higher score on the search for meaning items indicates greater active search for meaning. Maximum score: 70 Minimum score: 10.

OTHER OUTCOMES:
FACIT Spiritual Well-Being Scale | Pre-test (0 weeks) to Post-test (6 weeks)
  The spiritual well-being of RT-ALS dyads reported at baseline and post-test as measured by the FACIT Spiritual Well-Being scale. Maximum score: 4 Minimum score: 0 on each sub scale. Higher scores indicate higher spiritual well-being.
Concern with Dying Scale | Pre-test (0 weeks) to Post-test (6 weeks)
  Measure of concern with dying in RT-ALS dyads reported at baseline and post-test as measured by the Concern with Dying Scale. Maximum score: 20 Minimum score: 6. Higher scores indicate higher levels of concern with death and dying.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Rush, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No